CLINICAL TRIAL: NCT02265315
Title: Augmenting Treatment Effects of Voice Therapy in Parkinson Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Le Bonheur Children's Hospital (Other)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other); University of Tennessee (Other); University of Memphis (Other)
Responsible Party: Principal Investigator, James W. Wheless, Shalini Narayana, Ph.D., Le Bonheur Children's Hospital
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 14-03265-FB UM
Record Dates: First submitted 2014-10-09; First posted 2014-10-15 (Estimated); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- LSVT +sham TMS (Sham Comparator): Lee Silverman Voice Treatment (LSVT) and Transcranial Magnetic Stimulation (TMS)
  Interventions: Behavioral: Lee Silverman Voice Treatment
- LSVT +left rTMS (Active Comparator): Lee Silverman Voice Treatment (LSVT) and Transcranial Magnetic Stimulation (TMS) applied to left side of head
  Interventions: Other: Transcranial Magnetic Stimulation; Behavioral: Lee Silverman Voice Treatment
- LSVT + right rTMS (Active Comparator): Lee Silverman Voice Treatment (LSVT) and Transcranial Magnetic Stimulation (TMS) applied to right side of brain
  Interventions: Other: Transcranial Magnetic Stimulation; Behavioral: Lee Silverman Voice Treatment

INTERVENTIONS:
Other: Transcranial Magnetic Stimulation — Treament adjuvant applied to accelerate vocal motor learning and overall voice improvement
  Other Names: TMS
  Arms: LSVT + right rTMS; LSVT +left rTMS
Behavioral: Lee Silverman Voice Treatment — Time intensive behavioral treatment for Parkinson's hypophonia
  Other Names: LSVT

SUMMARY:
The purpose of this study is to evaluate the impact of a non-invasive brain stimulation technique called transcranial magnetic stimulation (TMS) on voice/speech treatment in people with Parkinson's Disease (PD), through the use of speech and voice analysis, examination of voice box, and brain imaging methods.

DETAILED DESCRIPTION:
Effective treatment of the speech disorder in IPD is as important as the optimal control of limb motor symptoms. Presently, the Lee Silverman Voice Treatment (LSVTÒ LOUD) - is a time intensive behavioral treatment for Parkinson's hypophonia. Facilitatory TMS is a safe and a complimentary stimulation technique. Brain imaging has also identified suitable target brain regions that are readily accessible to TMS. This combined treatment modality approach should be more effective and efficient the LSVT alone.

The study will enroll patients with Parkinson's disease with moderate to severe hypophonia. A total of 36 patients will be recruited over 3 years and divided into 3 groups (n=12 each). The three cohorts are: 1. LSVT +sham TMS; 2. LSVT +left rTMS and 3. LSVT + right rTMS.

This is a longitudinal double blind randomized controlled clinical trial. All investigators and study personnel will be blind to the study except for the PI responsible for TMS (Dr. Narayana). The entire protocol occurs over 19 weeks. During the first week, the participants will be screened, consented. During the second week, baseline behavioral and imaging data will be collected. Next, the patients will be randomized to one of the three treatment groups. Then the patients will enter a 4-week treatment phase, where they will receive TMS/sham TMS and LSVT 4 days a week for 4 weeks. During the seventh week, patients will undergo post treatment behavioral and imaging assessments. Then the patients will return in week 19 to complete the follow up behavioral measures and imaging session.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with Idiopathic Parkinson's disease (IPD) between the ages of 45 and 80 years with moderate to severe hypophonia
* None or mild cognitive impairment or depression
* Stable medication therapy for at least 3 months. Must be "optimally medicated" at the start of the study. This means that there should be no change in mediction type or dosage in 3 months prior to enrolling in the study. The medications should not be causing significant or serious advese effects

Exclusion Criteria:

* History of drug abuse or neurological condition other than or in addition to IPD (for example stroke)
* Individuals with advanced IPD (stage V) or who had LSVT within 3 years
* Pregnant females
* History of seizures, history of major head trauma, metal objects implanted in the head, ferrous metal filings in the eye, brain damage, inflammation of the brain, cardiac pacemaker, implanted medication pump, cardiac lines, heart disease, currently taking certain types of medication for depression or seizures (tricyclic antidepressants or neuroleptics which lower seizure threshold

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2014-10; Primary Completion 2020-12-31 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Clinical assessment: | 19 weeks
  Voice intensity and overall voice quality
Patient assessment: | 19 weeks
  10-item Voice related Quality of Life Scale (V-RQOL)
Physiological assessment: | 19 weeks
  Vocal fold function; Changes in brain activation: at the site of TMS stimulation and the speech motor network; and Functional connectivity within the speech motor network

SECONDARY OUTCOMES:
Clinical assessment | 19 weeks
  intelligibility and articulation
Patient self-assessment | 19 weeks
  visual analog scaling of speech intelligibility

CONTACTS AND LOCATIONS:
Overall Officials: Shalini Narayana, PhD, Principal Investigator — LeBonheur Children's Hospital
Locations (1):
- LeBonheur Children Hospital, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- See also: Michael J. Fox Trial Finder — https://foxtrialfinder.michaeljfox.org/trial/3885/